CLINICAL TRIAL: NCT03487250
Title: Prospective Multi-Center Evaluation of Percutaneous Ultrasound Guided Elbow Tenotomy (PUGET) Using the HydroCision TenJet HydroSurgery System
Brief Title: Percutaneous US Guided Elbow Tenotomy With the TenJet HydroSurgery System
Status: Completed | Type: Observational
Sponsor: HydroCision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PUGET-01-016
Record Dates: First submitted 2018-03-25; First posted 2018-04-03 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Elbow, Tennis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- TenJet System: Percutaneous ultrasound guided medial and lateral tenotomy using the TenJet HydroSurgery System
  Interventions: Device: TenJet System

INTERVENTIONS:
Device: TenJet System — Percutaneous ultrasound guided medial and lateral tenotomy using the TenJet HydroSurgery System

SUMMARY:
To evaluate the acute and long-term clinical outcomes of tenotomy with the TenJet System in patients with elbow tendinosis.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single arm post-marketing clinical study of patients undergoing percutaneous ultrasound guided medial and lateral tenotomy using the TenJet HydroSurgery System to treat elbow tendinosis. Patients will be followed for a maximum of 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years of age
* Chronic lateral or medial elbow pain > 3 month duration
* History and clinical examination consistent with lateral or medial epicondylitis
* Sonographic evidence of medial or lateral elbow tendinosis as evidenced by

  * tendon thickening and hypoechogenicity,
  * with or without hypervascularity on Doppler examination and,
  * with or without cortical irregularities, Or MRI findings consistent with lateral or medial tendinosis, with or without intrasubstance tear.
* > 3 months of non-operative treatment that included

  * nonsteroidal anti-inflammatory drugs
  * activity modification
  * physical therapy
  * elbow straps
  * With or without previous steroid injections, protein rich plasma injections, or stem cell injections
* Patient is willing and able to provide informed consent and comply with the study protocol

Exclusion Criteria:

* Documented ipsilateral upper extremity musculoskeletal condition (other than elbow tendinosis in the same arm on the opposite side)
* Bleeding disorders and/or current use of anti-coagulants with the inability to withhold anticoagulants for required time prior to procedure
* Use of acetylsalicylic acid (ASA) and/or non-steroidal anti-inflammatory drug (NSAID) within 7 days of treatment
* Steroid injection within 4 weeks of the study procedure
* Active local or systemic infection
* Patient found to have further degenerative changes of the elbow contributing to pain, such as cartilage thinning, loose body, or evidence of tendinosis other than medial or lateral, including triceps or ulnar collateral ligament.
* Patient is known or suspected to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic, refractory lateral or medial elbow pain secondary to elbow tendinosis
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Change in elbow pain using Visual Analog Scale (VAS) | Up to 12 months
  Change in elbow pain VAS compared to baseline

SECONDARY OUTCOMES:
Change in Elbow Function using the Patient-Rated Elbow Evaluation Questionnaire (PREE) | Up to 12 months
  Change in PREE compared to baseline
Pain medication usage | Up to 12 months
  Reduction in medications for elbow pain

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Kapteyn, DO, Principal Investigator — Orthopaedic Associates of Muskegon
Locations (3):
- United States (3):
  - Orthopaedic Associates of Muskegon, Muskegon, Michigan
  - Penn Highlands, DuBois, Pennsylvania
  - Noble Pain Management & Sports Medicine, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No